CLINICAL TRIAL: NCT01978626
Title: Enhancing Performance of Cognitive Behavioral Therapy for Insomnia With an Integrative Mobile Platform
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201307042RINC
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Primary Insomnia; Depressive Disorders With Insomnia
Keywords: Insomnia; Comorbid insomnia; Cognitive Behavioral Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smart phone Apps (Experimental): 1. 1st year: Electronic sleep diary module: an app with electronic sleep diary and message reminder
  2. 2nd year: Social persuasion system module: an app of smart phone that encourages participants with each others
  3. 3rd year: Tai-chi module: a multi-media oriented app that helps participants practice Tai-Chi
  Interventions: Behavioral: App modules
- Control (Active Comparator): 1. 1st year: traditional paper-pencil diary
  2. 2nd year: no social persuasion is given beyond sessions
  3. 3rd year: Tai-chi teaching by Digital Video Disc only
  Interventions: Behavioral: Traditional CBT-I

INTERVENTIONS:
Behavioral: App modules
  Arms: Smart phone Apps
Behavioral: Traditional CBT-I
  Arms: Control

SUMMARY:
Cognitive Behavioral Therapy for Insomnia (CBT-I) has been proven as an effective intervention for the non-pharmacological treatment of insomnia. This study hypothesizes app programs of smart phone would enhance the compliance and performance of behavioral intervention of CBT-I. During a 3-year study period, 3 app modules, including electronic sleep diary along with message reminder system, social persuasion system and Tai-Chi practice system will be tested subsequently for their efficacy.

DETAILED DESCRIPTION:
This study comprises 3 parts which are designed as an open-label, active-control study. In each year, the participants in the experimental arm receive app-assisted CBT-I. In the first year, participants with primary insomnia are recruited and assigned to the experimental arm or the active-control arm with matched age, gender and education status. The subject number in each arm is 20. Participants in each arm receive a 6-week standard CBT-I. In the experimental arm, the participants use electronic sleep diary and message reminder to record sleep pattern. In the active-control group, the participants use traditional paper-pencil sleep diary instead. In the second year, participants with primary insomnia are recruited and assigned to the experimental arm or the active-control arm with matched age, gender and education status. The subject number in each arm is 20. Participants in each arm receive a 6-week standard CBT-I. In the experimental arm, the participants use app with function of social persuasion to encourage each other. In the active-control group, no social persuasion is given beyond the treatment sessions. In the third year, participants with comorbid depressive disorder and insomnia are recruited and assigned to the experimental arm or the active-control arm with matched age, gender and education status. The subject number in each arm is 20. Participants in each arm receive a 6-week standard CBT-I. In the experimental arm, the participants use app module that provides a multi-media assisted Tai-Chi video to practice Tai-Chi. In the active-control group, a traditional Tai-CHi teaching digital video disc is provided to help the participants practice Tai-Chi.

ELIGIBILITY:
First and second year:

Inclusion criteria:

* 20 and more years old
* meet Diagnostic and Statistical Manual-IV diagnostic criteria for primary insomnia

Exclusion criteria:

* not current smart phone users

Third year:

Inclusion criteria:

* 20 and more years old
* meet Diagnostic and Statistical Manual-IV diagnostic criteria for depressive disorders (major depressive disorder or dysthymic disorder)
* mild to moderate severity of depression (Beck Depression Inventory: 13 and more but less than 29)
* mild anxiety symptoms (Bexk Anxiety Inventory: less than 10)

Exclusion criteria:

* with high suicide risk
* not current smart phone users

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of app on CBT-I (The first year) | 6 weeks
  The compliance rate of keeping sleep diary and behavioral prescription.
Efficacy of app on CBT-I (The second year) | 6 weeks
  The efficacy of social persuasion app module on sleep quality
Efficacy of app on CBT-I (The third year) | 6 weeks
  The efficacy of Tai-Chi multi-media app module on sleep quality

OTHER OUTCOMES:
Satisfaction on app | 6 weeks
  In the first year, the satisfaction of app design will be surveyed in the experimental arm.

CONTACTS AND LOCATIONS:
Overall Officials: Hsi-Chung Chen, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan